CLINICAL TRIAL: NCT00511797
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Comparative Study to Investigate the Optimal Dose of Drospirenone for Dysmenorrhea With SH T04740A [Drospirenone 1 mg/Ethinylestradiol 20 µg (as ß-cyclodextrin Clathrate)], SH T 04740E [Drospirenone 2 mg/Ethinylestradiol 20 µg (as ß-cyclodextrin Clathrate)] and SH T00186D [Drospirenone 3 mg/ Ethinylestradiol 20 µg (as ß-cyclodextrin Clathrate)] Administered Orally for 16 Weeks (4 Cycles), and to Confirm the Efficacy of SH T00186D for Dysmenorrhea.
Brief Title: SH T00186 Phase II/ III Optimal Drospirenone (DRSP) Dose Finding and Placebo-controlled Comparative Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91615; 310283 (Other: Company Internal)
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Results first posted 2010-10-04 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-11

CONDITIONS: Dysmenorrhea
Keywords: Dysmenorrhea; Dysmenorrheal score; Drospirenone; DRSP; Ethinylestradiol
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- DRSP 1 mg/EE 20 μg (Experimental): 1 tablet per day Drospirenone (DRSP) 1 mg/Ethinylestradiol (EE) 20 μg for 24 days and 1 tablet per day placebo for 4 days in each 28-day cycle
  Interventions: Drug: SH T04740B
- DRSP 2 mg/EE 20 μg (Experimental): 1 tablet per day Drospirenone (DRSP) 2 mg/Ethinylestradiol (EE) 20 μg for 24 days and 1 tablet per day placebo for 4 days in each 28-day cycle
  Interventions: Drug: SH T04740F
- DRSP 3 mg/EE 20 μg (Experimental): 1 tablet per day Drospirenone (DRSP) 3 mg/Ethinylestradiol (EE) 20 μg for 24 days and 1 tablet per day placebo for 4 days in each 28-day cycle
  Interventions: Drug: SH T00186DF
- Placebo (Placebo Comparator): 1 tablet per day placebo for 28 days in each 28-day cycle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SH T04740B — Drospirenone 1mg/EE 20µg (ß-CDC)
  Arms: DRSP 1 mg/EE 20 μg
Drug: SH T00186DF — Drospirenone 3 mg/EE 20µg (ß-CDC)
  Arms: DRSP 3 mg/EE 20 μg
Drug: SH T04740F — Drospirenone 2 mg/EE 20µg (ß-CDC)
  Arms: DRSP 2 mg/EE 20 μg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate efficacy of drospirenone for dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years or older at obtaining informed consent
* Patients having the normal menstrual cycle (28+/-3 days) in the latest two menses before the final enrollment
* Patients having a total dysmenorrhea score of at least 3 points in two menstrual cycles before the final enrollment

Exclusion Criteria:

* Patients with ovarian chocolate cysts and symptomatic uterine fibroids (as defined in greater detail in the study protocol)
* Patients with estrogen-dependent tumors (e.g. breast cancer, cancer of the uterine body or breast fibrocystic, etc.), and patients with cervical cancer or suspected cervical cancer (e.g. class III or greater in the cervical smear or endometrial smear examination.)
* Patients with undiagnosed abnormal vaginal bleeding
* Patients with thrombophlebitis, pulmonary embolism, cerebrovascular disease(including transient ischemic attack, etc.), or coronary artery disease(e.g. myocardial infarction and angina pectoris, etc.), or a history of those diseases
* Patients aged 35 years or older who smoke at least 15 cigarettes per day
* Patients with migraine accompanied by prodrome (e.g. scintillating scotoma or star-shaped scintillation)
* Patients with pulmonary hypertension or valvular heart disease complicated by atrial fibrillation, and patients with a history of subacute bacterial endocarditis
* Patients who are regularly taking nutritional products that contain St. John's Wort
* Patients who underwent surgical treatment for endometriosis by laparotomy, or laparoscopy within 2 months prior to screening
* Patients who need to use analgesics regularly for therapeutic objectives other than relief from the pain of dysmenorrhea during this study (occasional use permitted)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- Japan (11):
  - Maebashi, Gunma
  - Kobe, Hyōgo
  - Nishinomiya, Hyōgo
  - Yokohama, Kanagawa
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Osaka, Osaka
  - Chuo-ku, Tokyo
  - Hachiōji, Tokyo
  - Setagaya-ku, Tokyo
  - Toshima-ku, Tokyo

REFERENCES:
- [Result] Momoeda M, et al. Treatment of Functional and Organic Dysmenorrhea - Investigation of the Efficacy and Safety of Drospirenone/Ethinylestradiol Combination Tablet (YAZ). Sanka to Fujinka (Obstetrics and Gynecology), 2010: 77 (8) 977-88 (in Japanese)
- [Derived] Schroll JB, Black AY, Farquhar C, Chen I. Combined oral contraceptive pill for primary dysmenorrhoea. Cochrane Database Syst Rev. 2023 Jul 31;7(7):CD002120. doi: 10.1002/14651858.CD002120.pub4. PMID 37523477

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Full Analysis Set (FAS) consisted of all patients who received at least one dose of study drug. Patients were analyzed as treated.
  FAS was the primary analysis set for all efficacy endpoints and safety analyses. Per Protocol Set (PPS) was a subgroup of the FAS. The PPS consisted of patients in the FAS who did not have major protocol deviations.
Period: Overall Study
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Started | 62 | 63 | 62 | 62
Subjects Dispensed Drugs | 61 | 63 | 61 | 59
Subjects Received Treatment | 61 (FAS) | 62 (FAS) | 61 (FAS) | 58 (FAS)
Completed | 55 | 55 | 51 | 47
Not Completed | 7 | 8 | 11 | 15
Not completed — Adverse Event | 1 | 2 | 2 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 2 | 2 | 3
Not completed — Withdrawal by Subject | 3 | 3 | 4 | 2
Not completed — Never dispensed | 1 | 0 | 1 | 3
Not completed — Study drug not taken | 0 | 1 | 0 | 1
Not completed — Partially missing diary | 0 | 0 | 1 | 0
Not completed — Other (moving etc) | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo | Total
Number analyzed (Participants) | 61 | 62 | 61 | 58 | 242
Age, Continuous [Mean (Full Range); unit: years] | 31.0 [21 to 45] | 30.6 [20 to 43] | 30.9 [20 to 48] | 30.8 [20 to 44] | 30.8 [20 to 48]
Gender [Count of Participants; unit: Participants]
  Female | 61 | 62 | 61 | 58 | 242
  Male | 0 | 0 | 0 | 0 | 0
Diagnosis type [Number; unit: participants]
  Functional dysmenorrhea | 47 | 48 | 42 | 41 | 178
  Organic dysmenorrhea | 14 | 14 | 19 | 17 | 64
Details of organic dysmenorrhea [Number; unit: participants] — Not all participants had organic dysmenorrhea. Some of participants were diagnosed as having a multiple type of organic dysmenorrhea.
  participants
    Endometriosis | 1 | 3 | 4 | 5 | 13
    Uterine fibroids | 9 | 7 | 10 | 9 | 35
    Uterine adenomyosis | 6 | 7 | 11 | 8 | 32
    Bicornuate uterus | 2 | 0 | 0 | 0 | 2
Average length of menstrual cycle [Mean (Full Range); unit: days] | 28.6 [25 to 31] | 28.7 [25 to 33] | 28.3 [25 to 32] | 28.7 [25 to 31] | 28.6 [25 to 33]
Body mass index (BMI) [Mean (Full Range); unit: kg/m^2] | 21.05 [15.6 to 30.0] | 20.41 [16.6 to 25.8] | 20.67 [16.4 to 29.9] | 21.19 [17.2 to 27.7] | 20.82 [15.6 to 30.0]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Dysmenorrheal Score at Final Evaluation
Description: Total dysmenorrheal score was defined as sum of 2 sub-scores: severity of dysmenorrhea (none: 0, mild: 1, moderate: 2, severe: 3) and use of analgesics (none: 0, mild: 1, moderate: 2, severe: 3). Total possible best is 0, and total possible worst is 6. Note: used with permission of Nobelpharma Co., Ltd. from the phase 3 clinical study protocol (Prog Med 2005:25 (3):739-758) of IKH-01 in dysmenorrhea (associated with endometriosis) (Nobelpharma Co., Ltd.)
Time Frame: Baseline and up to 4 Cycles (28 days per cycle)
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 61 | 62 | 61 | 58
scores on a scale | -2.5 (1.52) | -2.1 (1.51) | -1.9 (1.63) | -1.0 (1.53)
Statistical Analysis 1: Comparison: DRSP 3 mg/EE 20 μg vs Placebo; Three null hypotheses were sequentially tested. H01: DRSP 3 mg >= Placebo (Active is equal or less in decrease of score) vs H11: DRSP 3 mg < Placebo (Active is greater in decrease of score), H02: DRSP 2 mg >= Placebo vs H12: DRSP 2 mg < Placebo, H03: DRSP 1 mg >= Placebo vs H13: DRSP 1 mg < Placebo; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Pre-defined sequential tests were applied to protect alpha inflation by multiplicity; Median Difference (Final Values) = -0.92, 95% CI 2-sided [-1.49 to -0.34], Standard Error of Mean 0.290
Statistical Analysis 2: Comparison: DRSP 2 mg/EE 20 μg vs Placebo; Second null hypothesis was tested. H02: DRSP 2 mg >= Placebo vs H12: DRSP 2 mg < Placebo; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; Median Difference (Final Values) = -1.10, 95% CI [-1.64 to -0.55], Standard Error of Mean 0.277
Statistical Analysis 3: Comparison: DRSP 1 mg/EE 20 μg vs Placebo; Third null hypotheses was tested. H03: DRSP 1 mg >= Placebo vs H13: DRSP 1 mg < Placebo; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; Median Difference (Final Values) = -1.44, 95% CI [-2.00 to -0.89], Standard Error of Mean 0.280

2. Secondary Outcome: Change From Baseline in Total Dysmenorrheal Score at Cycle 1 up to Cycle 4
Description: Total dysmenorrheal score was defined as sum of 2 sub-scores: severity of dysmenorrhea (none: 0, mild: 1, moderate: 2, severe: 3) and use of analgesics (none: 0, mild: 1, moderate: 2, severe: 3). Total possible best is 0, and total possible worst is 6.
Time Frame: Baseline and up to 4 Cycles (28 days per cycle)
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 61 | 62 | 61 | 58
scores on a scale
  Cycle 1 | -2.4 (1.40) | -2.1 (1.49) | -1.8 (1.67) | -0.8 (1.50)
  Cycle 2 | -2.1 (1.40) | -2.3 (1.57) | -1.9 (1.50) | -1.1 (1.59)
  Cycle 3 | -2.5 (1.34) | -2.3 (1.52) | -2.1 (1.34) | -1.0 (1.59)
  Cycle 4 | -2.5 (1.55) | -2.3 (1.41) | -2.1 (1.54) | -1.0 (1.63)
Statistical Analysis 1: Comparison: DRSP 3 mg/EE 20 μg vs Placebo; Test results of 3 mg DRSP and placebo at Cycle 4 are shown. 2-sided 95% confidence intervals were calculated. To keep consistency with 2-sided 95% confidence intervals, 2.5% 1-sided significance levels were used for the statistical tests; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-1.74 to -0.46], Standard Error of Mean 0.322
Statistical Analysis 2: Comparison: DRSP 2 mg/EE 20 μg vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = -1.34, 95% CI [-1.95 to -0.73], Standard Error of Mean 0.306
Statistical Analysis 3: Comparison: DRSP 1 mg/EE 20 μg vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = -1.53, 95% CI [-2.16 to -0.90], Standard Error of Mean 0.317

3. Secondary Outcome: Number of Participants With Severity of Lower Abdominal Pain During Menstruation at Cycle 4
Description: Severity of lower abdominal pain during menstruation was rated as none (none), mild (can be easily tolerated), moderate (noticeable, but does not interfere with daily activities), or severe (interferes with daily activities).
Time Frame: Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Number; unit: participants
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 55 | 53 | 51 | 46
participants
  none | 15 | 17 | 11 | 3
  mild | 28 | 27 | 19 | 11
  moderate | 9 | 7 | 14 | 21
  severe | 3 | 2 | 7 | 11

4. Secondary Outcome: Number of Participants With Severity of Low Back Pain During Menstruation at Cycle 4
Description: Severity of low back pain during menstruation was rated as none (none), mild (can be easily tolerated), moderate (noticeable, but does not interfere with daily activities), or severe (interferes with daily activities).
Time Frame: Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Number; unit: participants
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 55 | 53 | 51 | 46
participants
  none | 34 | 36 | 30 | 18
  mild | 15 | 12 | 18 | 14
  moderate | 5 | 4 | 2 | 9
  severe | 1 | 1 | 1 | 5

5. Secondary Outcome: Number of Participants With Severity of Headache During Menstruation at Cycle 4
Description: Severity of headache during menstruation was rated as none (none), mild (can be easily tolerated), moderate (noticeable, but does not interfere with daily activities), or severe (interferes with daily activities).
Time Frame: Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Number; unit: participants
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 55 | 53 | 51 | 46
participants
  none | 47 | 35 | 39 | 29
  mild | 5 | 10 | 5 | 6
  moderate | 1 | 6 | 3 | 6
  severe | 2 | 2 | 4 | 5

6. Secondary Outcome: Number of Participants With Severity of Nausea or Vomiting During Menstruation at Cycle 4
Description: Severity of nausea or vomiting during menstruation was rated as none (none), mild (can be easily tolerated), moderate (noticeable, but does not interfere with daily activities), or severe (interferes with daily activities).
Time Frame: Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Number; unit: participants
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 55 | 53 | 51 | 46
participants
  none | 51 | 47 | 47 | 40
  mild | 2 | 4 | 4 | 4
  moderate | 2 | 1 | 0 | 2
  severe | 0 | 1 | 0 | 0

7. Secondary Outcome: Number of Participants With Total Pelvic Pain Score at Times Other Than During Menstruation at Cycle 4
Description: Total pelvic pain score was defined as sum of 2 sub-scores: severity of dysmenorrhea and use of analgesics. Higher score means it is more severe. 0=None, 6=Severest.
Time Frame: Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Number; unit: participants
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 55 | 53 | 51 | 46
participants
  0 | 40 | 41 | 42 | 30
  1 | 11 | 10 | 7 | 6
  2 | 3 | 2 | 1 | 5
  3 | 0 | 0 | 0 | 3
  4 | 0 | 0 | 0 | 1
  5 | 1 | 0 | 1 | 1
  6 | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) for Dysmenorrhea at Times Other Than During Menstruation at Cycle 4
Description: VAS is an unmarked scale on a line 100 mm in length, indicating from 0 mm (no pain) to 100 mm (worst pain a participant has ever experienced).
Time Frame: From baseline up to Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 55 | 53 | 51 | 46
scores on a scale | -43.0 (23.44) | -39.5 (22.12) | -31.8 (23.55) | -10.3 (24.53)

9. Secondary Outcome: Visual Analogue Scale (VAS) for Pelvic Pain at Times Other Than During Menstruation at Cycle 4
Description: as for outcome 8
Time Frame: Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 55 | 53 | 51 | 46
scores on a scale | 5.9 (11.52) | 5.4 (11.78) | 4.0 (14.26) | 11.5 (20.22)

10. Secondary Outcome: Change From Baseline in Endometrial Thickness After 4-cycle Treatment
Description: Endometrial thickness was measured via transvaginal ultrasound examination. The endometrium is the inner membrane of the uterus. During the menstrual cycle, the endometrium grows to a thick, blood vessel-rich, glandular tissue layer.
Time Frame: From baseline to Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 53 | 53 | 50 | 47
mm | -5.5 (4.11) | -7.1 (3.25) | -6.3 (4.07) | -0.1 (2.79)

11. Secondary Outcome: Number of Bleeding / Spotting Episodes
Description: Bleeding data were captured from the diary a participant recorded by herself. Bleeding is a genital bleeding. Spotting is a slight genital bleeding with participant's experience. An episode means a series of bleeding and/or spotting. The bleeding /spotting analyses are by intensity.
Time Frame: For the first 90 days
Population: FAS (Participants with the defined data)
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 59 | 60 | 57 | 56
number of episodes
  bleeding / spotting | 3.3 (0.9) | 3.3 (1.3) | 3.4 (0.9) | 2.9 (0.9)
  bleeding only | 0.5 (0.9) | 0.4 (0.8) | 0.3 (0.5) | 0.4 (0.8)
  spotting only | 0.3 (0.6) | 0.4 (1.1) | 0.4 (0.8) | 0.2 (0.6)

12. Secondary Outcome: Number of Bleeding / Spotting Days
Description: Bleeding data were captured from the diary a participant recorded by herself. Bleeding is a genital bleeding. Spotting is a slight genital bleeding with participant's experience. The bleeding /spotting analyses are by intensity.
Time Frame: For the first 90 days
Population: FAS (Participants with the defined data)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 59 | 60 | 57 | 56
days
  bleeding / spotting | 32.3 (8.7) | 31.2 (11.4) | 29.2 (11.0) | 22.6 (5.5)
  bleeding only | 21.3 (5.9) | 19.3 (8.8) | 18.6 (6.5) | 17.4 (4.9)
  spotting only | 11.1 (7.0) | 11.9 (7.6) | 10.5 (8.2) | 5.2 (2.5)

13. Secondary Outcome: Participants With Withdrawal Bleeding
Description: Withdrawal bleedings were defined as bleedings while a participant takes placebo tablets.
Time Frame: At Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Number; unit: participants
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 55 | 55 | 52 | 48
participants | 50 | 50 | 49 | 47

14. Secondary Outcome: Participants With Intracyclic Bleeding
Description: Intracyclic bleedings were defined as bleedings while a participant takes active drugs.
Time Frame: At Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Number; unit: participants
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 55 | 55 | 52 | 48
participants | 14 | 8 | 8 | 4

15. Secondary Outcome: Participants With Non-heavy Intracyclic Bleeding
Description: Non-heavy bleedings were defined as those other than heavy bleeding (less or normal bleeding).
Time Frame: At Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Number; unit: participants
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 14 | 8 | 8 | 4
participants | 14 | 8 | 7 | 2

16. Secondary Outcome: Participants With Non-heavy Withdrawal Bleeding
Description: Non-heavy bleedings were defined as those other than heavy bleeding (less or normal bleeding).
Time Frame: At Cycle 4 (28 dyas per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Number; unit: participants
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 50 | 50 | 49 | 47
participants | 45 | 44 | 42 | 38

17. Secondary Outcome: Change From Baseline in Serum Carbohydrate Antigen-125 (CA125) After 4-cycle Treatment
Description: CA125 is a laboratory parameter giving an indication of having tumor, whose elevated levels that were defined by a lab suggest a potential tumor.
Time Frame: From baseline to Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Mean (Full Range); unit: Units/L
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 55 | 55 | 51 | 47
Units/L | -2.78 [-26.4 to 5.5] | 0.53 [-17.4 to 184.9] | -3.79 [-35.6 to 32.5] | 0.89 [-7.8 to 15.8]

18. Secondary Outcome: Change From Baseline in Serum C-reactive Protein (CRP) After 4-cycle Treatment
Description: CRP is a laboratory parameter giving an indication of inflammation, whose elevated levels that were defined by a lab suggest a potential inflammation.
Time Frame: From baseline to Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 55 | 55 | 51 | 47
mg/dL | 0.015 [-0.31 to 0.85] | 0.042 [-0.09 to 0.77] | -0.014 [-2.73 to 0.35] | -0.175 [-7.38 to 0.62]

19. Secondary Outcome: Change From Baseline in Serum Estradiol Level After 4-cycle Treatment
Description: Estradiol is a predominant sex hormone that presents in female.
Time Frame: From baseline to Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 55 | 55 | 51 | 48
pg/mL | -18.32 [-341.5 to 968.9] | -42.23 [-336.8 to 329.0] | -98.02 [-477.8 to 231.2] | 49.20 [-182.7 to 310.3]

20. Secondary Outcome: Change From Baseline in Serum Progesterone Level at Cycle 4
Description: Progesterone is a steroid hormone involving in the female menstrual cycle, pregnancy, etc.
Time Frame: From baseline to Cycle 4 (28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 54 | 53 | 50 | 47
ng/mL | -7.93 [-22.2 to 6.3] | -8.23 [-23.6 to 5.7] | -9.37 [-22.3 to 6.7] | -0.27 [-20.6 to 18.7]

21. Post Hoc Outcome: Change From Baseline for Total Pelvic Pain Score at Times Other Than During Menstruation at Cycle 4
Description: Total pelvic pain score was defined as sum of 2 sub-scores: severity of dysmenorrhea (none: 0, mild: 1, moderate: 2, severe: 3) and use of analgesics (none: 0, mild: 1, moderate: 2, severe: 3). Total possible best is 0, and total possible worst is 6.
Time Frame: From baseline to Cycle 4(28 days per cycle)
Population: FAS (Participants with data at Cycle 4)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 55 | 53 | 51 | 46
scores on a scale | -0.1 (1.19) | -0.3 (1.12) | -0.1 (1.06) | 0.1 (1.22)

22. Post Hoc Outcome: Change From Baseline in Total Dysmenorrheal Score at Final Evaluation in Subgroups (1)
Description: as for outcome 1
Time Frame: Baseline and up to Cycle 4 (28 days per cycle)
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 61 | 62 | 61 | 58
scores on a scale
  age: < 30 years | -2.2 (1.46) | -2.4 (1.50) | -1.9 (1.49) | -1.2 (1.45)
  age: >= 30 years | -2.8 (1.54) | -1.9 (1.49) | -1.9 (1.75) | -0.8 (1.60)
  weight: < 50 kg | -3.0 (1.30) | -2.4 (0.99) | -1.5 (1.39) | -0.7 (1.65)
  weight: >= 50kg | -2.1 (1.57) | -2.0 (1.64) | -2.2 (1.74) | -1.1 (1.50)
  functional dysmenorrhea | -2.3 (1.63) | -2.1 (1.52) | -1.8 (1.73) | -1.0 (1.47)
  organic dysmenorrhea | -2.9 (1.00) | -2.1 (1.49) | -2.3 (1.37) | -1.0 (1.70)
  with medical surgical history | -2.3 (1.62) | -2.0 (1.50) | -2.1 (1.61) | -1.1 (1.68)
  without medical surgical history | -2.6 (1.42) | -2.3 (1.53) | -1.8 (1.66) | -0.8 (1.27)

23. Post Hoc Outcome: Change From Baseline in Total Dysmenorrheal Score at Final Evaluation in Subgroups (2)
Description: as for outcome 1
Time Frame: Baseline and up to 4 Cycles (28 days per cycle)
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 61 | 62 | 61 | 58
scores on a scale
  with previous medication | -2.5 (1.53) | -2.1 (1.51) | -1.9 (1.63) | -1.0 (1.53)
  with pregnancy history | -2.7 (1.62) | -1.9 (1.32) | -2.2 (1.72) | -1.0 (2.03)
  without pregnancy history | -2.3 (1.47) | -2.2 (1.62) | -1.8 (1.61) | -1.0 (1.22)
  with birth history | -2.9 (1.59) | -2.1 (1.28) | -2.3 (1.96) | -1.1 (2.00)
  without birth history | -2.3 (1.49) | -2.1 (1.62) | -1.9 (1.55) | -1.0 (1.35)
  total dysmenorrheal score at baseline: 3 or 4 | -2.1 (1.28) | -1.9 (1.36) | -1.8 (1.44) | -1.0 (1.49)
  total dysmenorrheal score at baseline: 5 or 6 | -3.4 (1.75) | -2.6 (1.77) | -2.4 (2.06) | -1.1 (1.65)

24. Post Hoc Outcome: Change From Baseline in Total Dysmenorrheal Score at Final Evaluation in Patients Without Previous Medication
Description: as for outcome 1
Time Frame: Baseline and up to 4 Cycles (28 days per cycle)
Population: The number of subjects without previous medication in DRSP 1 mg/EE 20 μg group was 1, so the standard deviation was not measurable. The number of subjects without previous medication in the other three groups were 0, so the data were not applicable.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Number analyzed (Participants) | 1 | 0 | 0 | 0
scores on a scale | -2.0 |  |  |

ADVERSE EVENTS:
Arm/Group | DRSP 1 mg/EE 20 μg | DRSP 2 mg/EE 20 μg | DRSP 3 mg/EE 20 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/62 | 2/63 | 0/62 | 1/62
Other Adverse Events (participants affected / at risk) | 56/62 | 58/63 | 60/62 | 53/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DRSP 1 mg/EE 20 μg (N=62) | DRSP 2 mg/EE 20 μg (N=63) | DRSP 3 mg/EE 20 μg (N=62) | Placebo (N=62)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DRSP 1 mg/EE 20 μg (N=62) | DRSP 2 mg/EE 20 μg (N=63) | DRSP 3 mg/EE 20 μg (N=62) | Placebo (N=62)
Abdominal pain lower (Gastrointestinal disorders) | 5 (5) | 7 (10) | 9 (10) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (6) | 5 (6) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (10) | 3 (3) | 4 (4)
Blood triglycerides increased (Investigations) | 5 (5) | 1 (1) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (2) | 3 (3) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 5 (7) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 16 (30) | 18 (26) | 22 (47) | 26 (58)
Headache (Nervous system disorders) | 21 (48) | 28 (84) | 30 (63) | 23 (68)
Malaise (General disorders) | 2 (3) | 4 (4) | 3 (4) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 20 (34) | 18 (32) | 8 (12) | 4 (7)
Nasopharyngitis (Infections and infestations) | 17 (24) | 24 (35) | 24 (32) | 26 (32)
Nausea (Gastrointestinal disorders) | 16 (28) | 18 (32) | 22 (31) | 17 (30)
Prothrombin time shortened (Investigations) | 0 (0) | 2 (2) | 0 (0) | 4 (6)
Seasonal allergy (Immune system disorders) | 4 (5) | 2 (2) | 4 (4) | 5 (5)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 4 (4) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 8 (8) | 8 (8) | 8 (9) | 8 (8)
Genital haemorrhage (Reproductive system and breast disorders) | 20 (32) | 19 (31) | 23 (33) | 8 (8)
Coagulation test abnormal (Investigations) | 9 (9) | 6 (6) | 13 (13) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor will confirm the contents before disclosure.